CLINICAL TRIAL: NCT03766165
Title: The Engaging Microenterprise for Resource Generation and Health Empowerment (EMERGE) Project: Feasibility Trial of an Enhanced Microenterprise Intervention to Reduce Sexual Risk Behaviors in Young Adults
Brief Title: Microenterprise Intervention to Reduce Sexual Risk Behaviors in Young Adults
Acronym: EMERGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00008833; K01MH107310 (NIH)
Record Dates: First submitted 2018-12-04; First posted 2018-12-06 (Actual); Results first posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-09

CONDITIONS: Feasibility
MeSH Terms: interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Job announcements plus educational sessions, mentoring, behavioral economic text messages, and a start-up grant.
  Interventions: Behavioral: Intervention
- Control (Other): Job announcements only
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Intervention — Participants will receive job announcements plus educational sessions, mentoring, behavioral economic text messages, and a start-up grant.
  Arms: Intervention
Behavioral: Control — Participants will receive job announcements only.
  Arms: Control

SUMMARY:
The study team will conduct a two-group study to examine the feasibility of implementing an enhanced microenterprise intervention to reduce sexual risk behaviors. The team will enroll approximately 40 young adults. Participants will be randomly assigned to one of two groups. The first group ("control") will receive text messages with information on job openings. The second group ("intervention") will receive text messages with information on job openings plus HIV prevention and business educational sessions, mentored apprenticeship, a start-up grant (provided in 6 payments), and HIV behavioral economics text messages.

DETAILED DESCRIPTION:
The study team will conduct a two-group study to examine the feasibility of implementing an enhanced microenterprise intervention to reduce sexual risk behaviors. The team will enroll approximately 40 young adults, aged 18 to 24, who are African-American, homeless, out-of-school, unemployed or under-employed, report unprotected/unsafe sex, and have access to a cell phone. Participants will be randomly assigned to one of two groups. The first group ("control") will receive text messages with information on job openings. The second group ("intervention") will receive text messages with information on job openings plus HIV prevention and business educational sessions, mentored apprenticeship, a start-up grant (provided in 6 payments), and HIV behavioral economics text messages. Data will be collected for 26 weeks (week 1 to week 26). Participants will undergo a baseline in-person interview at the time of enrollment (week 1) and be randomized to a group after completing a 3-week run-in period (week 1 to week 3). Each group will receive the assigned activities for 20 weeks (week 4 to week 23). An endline in-person interview will be conducted in and around week 26, respectively. Participants will also complete a weekly text message survey from enrollment (week 1) to the end of the study (week 26). The study team will collect feasibility information pertaining to two primary outcomes: (i) the proportion of participants in both groups who have responded to 70% or more of the weekly text message surveys at week 26 and (ii) the proportion of participants in the intervention group who have completed 70% or more of intervention activities (i.e., text message receipt, session attendance, grant spending, and mentor contact) at week 23. As secondary outcomes, the study team will collect feasibility information about the proportion of all participants who receive one or more informational text messages each week, the proportion of all participants who respond to a text message survey each week, the proportion of intervention participants who attend an educational session each week, the proportion of intervention participants who receive one or more mentor contacts each week, and the proportion of intervention participants who spend one or more grant payments each week. The study team will also examine the completion and variation in behavioral outcomes pertaining to the proportion of participants in each group who report one or more unprotected/unsafe sex acts in the last week and last month, the proportion of participants in each group who report one or more safer sex acts in the last week and last month, the proportion of participants in each group who report one or more HIV prevention care-seeking or information-seeking acts in the last week and last month, and the proportion of participants in each group who report one or more paid hours of work in the last week and last month. The study is anticipated to start in December 2018.

ELIGIBILITY:
Inclusion criteria are:

* African American;
* Aged 18-24;
* Living in Baltimore City;
* Having experienced one episode of homelessness in last 12 months;
* Unemployed or employed fewer than 10 hours per week;
* Not enrolled in school;
* Owning a mobile phone with text messaging function;
* Reporting at least one episode of unprotected/unsafe sex in prior 12 months

Exclusion criteria are:

* Aged 17 or younger;
* Older than 24 years;
* Unwilling to provide consent for study participation

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2019-08-19 (Actual); Study Completion 2019-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larissa Jennings Mayo-Wilson, PhD MHS, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data (IPD) will be shared.
Supporting Information: Study Protocol
Time Frame: The IPD will be posted on a permanent online data repository within 36 months after study completion.
Access Criteria: There are no access criteria.

REFERENCES:
- [Derived] Jennings Mayo-Wilson L, Coleman J, Timbo F, Latkin C, Torres Brown ER, Butler AI, Conserve DF, Glass NE. Acceptability of a feasibility randomized clinical trial of a microenterprise intervention to reduce sexual risk behaviors and increase employment and HIV preventive practices (EMERGE) in young adults: a mixed methods assessment. BMC Public Health. 2020 Dec 2;20(1):1846. doi: 10.1186/s12889-020-09904-x. PMID 33267860
- [Derived] Jennings Mayo-Wilson L, Coleman J, Timbo F, Ssewamala FM, Linnemayr S, Yi GT, Kang BA, Johnson MW, Yenokyan G, Dodge B, Glass NE. Microenterprise Intervention to Reduce Sexual Risk Behaviors and Increase Employment and HIV Preventive Practices Among Economically-Vulnerable African-American Young Adults (EMERGE): A Feasibility Randomized Clinical Trial. AIDS Behav. 2020 Dec;24(12):3545-3561. doi: 10.1007/s10461-020-02931-0. PMID 32494942
- [Derived] Mayo-Wilson LJ, Glass NE, Ssewamala FM, Linnemayr S, Coleman J, Timbo F, Johnson MW, Davoust M, Labrique A, Yenokyan G, Dodge B, Latkin C. Microenterprise intervention to reduce sexual risk behaviors and increase employment and HIV preventive practices in economically-vulnerable African-American young adults (EMERGE): protocol for a feasibility randomized clinical trial. Trials. 2019 Jul 17;20(1):439. doi: 10.1186/s13063-019-3529-7. PMID 31315685

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Control
Started | 19 | 19
Completed | 19 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Continuous [Mean (Full Range); unit: Years] | 21 [18 to 24] | 21 [18 to 24] | 21 [18 to 24]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 6 | 7 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 19 | 38
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 19 | 38
One or more episodes of homelessness within last 12 months [Count of Participants; unit: Participants] | 19 | 19 | 38

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants in Both Groups Who Have Responded to 70% or More of the Weekly Text Message Surveys
Description: Proportion of participants in both groups who have responded to 70% or more of the weekly text message surveys (description)
Time Frame: Measured at week 26
Population: Participants in both groups
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 19 | 19
Participants | 5 | 9

2. Primary Outcome: Proportion of Intervention Participants Who Have Completed 70% or More of Intervention Activities (i.e., Text Message Receipt, Session Attendance, Grant Spending, and Mentor Contact)
Description: Proportion of intervention participants who have completed 70% or more of intervention activities (i.e., text message receipt, session attendance, grant spending, and mentor contact) (description)
Time Frame: Measured at week 23
Population: Intervention participants
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 19
Participants | 11

3. Secondary Outcome: Proportion of All Participants Who Receive One or More Informational Text Messages
Description: Proportion of all participants who receive one or more informational text messages (description)
Time Frame: Measured weekly at week 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, and 23
Population: All participants
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: All participants including those in intervention arm and control arm
Arm/Group | All Participants
Number analyzed (Participants) | 38
Participants
  Week 4 | 38
  Week 5 | 38
  Week 6 | 38
  Week 7 | 38
  Week 8 | 38
  Week 9 | 38
  Week 10 | 38
  Week 11 | 38
  Week 12 | 38
  Week 13 | 38
  Week 14 | 38
  Week 15 | 38
  Week 16 | 38
  Week 17 | 38
  Week 18 | 38
  Week 19 | 38
  Week 20 | 37

4. Secondary Outcome: Proportion of All Participants Who Respond to the Text Message Survey
Description: Proportion of all participants who respond to the text message survey (description)
Time Frame: Measured weekly at week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24, 25, and 26
Population: All participants including those in intervention arm and control arm
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 38
Participants
  Week 1 | 29
  Week 2 | 33
  Week 3 | 34
  Week 4 | 31
  Week 5 | 31
  Week 6 | 29
  Week 7 | 28
  Week 8 | 23
  Week 9 | 22
  Week 10 | 25
  Week 11 | 25
  Week 12 | 23
  Week 13 | 23
  Week 14 | 23
  Week 15 | 23
  Week 16 | 23
  Week 17 | 18
  Week 18 | 16
  Week 19 | 16
  Week 20 | 15
  Week 21 | 14
  Week 22 | 15
  Week 23 | 17
  Week 24 | 16
  Week 25 | 17
  Week 26 | 14

5. Secondary Outcome: Proportion of Intervention Participants Who Attend an Educational Session
Description: Proportion of intervention participants who attend an educational session (description)
Time Frame: Measured weekly at week 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, and 23
Population: Intervention Participants Allowed on Site by CBO
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 17
Participants
  Week 4 | 12
  Week 5 | 12
  Week 6 | 12
  Week 7 | 10
  Week 8 | 11
  Week 9 | 10
  Week 10 | 11
  Week 11 | 10
  Week 12 | 11
  Week 13 | 8
  Week 14 | 8
  Week 15 | 7
  Week 16 | 6
  Week 17 | 5
  Week 18 | 5
  Week 19 | 3
  Week 20 | 3
  Week 21 | 4
  Week 22 | 4
  Week 23 | 6

6. Secondary Outcome: Proportion of Intervention Participants Who Receive One or More Mentor Contacts
Description: Proportion of intervention participants who receive one or more mentor contacts (description)
Time Frame: Measured weekly at week 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, and 23
Population: Intervention Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 19
Participants
  Week 4 | 0
  Week 5 | 0
  Week 6 | 0
  Week 7 | 0
  Week 8 | 0
  Week 9 | 11
  Week 10 | 11
  Week 11 | 8
  Week 12 | 4
  Week 13 | 7
  Week 14 | 3
  Week 15 | 4
  Week 16 | 2
  Week 17 | 2
  Week 18 | 5
  Week 19 | 4
  Week 20 | 3
  Week 21 | 2
  Week 22 | 2
  Week 23 | 2

7. Secondary Outcome: Proportion of Intervention Participants Who Spend One or More Grant Payments
Description: Proportion of intervention participants who spend one or more grant payments (description)
Time Frame: Measured weekly at week 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, and 23
Population: Intervention participants
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 19
Participants
  Week 4 | 0
  Week 5 | 0
  Week 6 | 0
  Week 7 | 0
  Week 8 | 0
  Week 9 | 0
  Week 10 | 11
  Week 11 | 11
  Week 12 | 11
  Week 13 | 11
  Week 14 | 11
  Week 15 | 11
  Week 16 | 11
  Week 17 | 6
  Week 18 | 6
  Week 19 | 6
  Week 20 | 5
  Week 21 | 5
  Week 22 | 5
  Week 23 | 5

8. Secondary Outcome: Proportion of Participants in Each Group Who Report One or More Unprotected Sex Acts in Last Week
Description: Proportion of participants in each group who report one or more unprotected sex acts in last week (description)
Time Frame: as for outcome 4
Population: Outcomes 8, 10, 12, 14 were collected using experimental text messages. As specified, if not feasible, an in-person pre- and post-intervention paper questionnaire would be used and report via Outcomes 9, 11, 13, 15 that are identical to Outcomes 8, 10, 12, 14, respectively. Text messages require modifications given high missing and accurate data.
Arm/Group | All Participants
Number analyzed (Participants) | 0

9. Secondary Outcome: Proportion of Participants in Each Group Who Report One or More Unprotected Sex Acts in Last Month
Description: Proportion of participants in each group who report one or more unprotected sex acts in last month (description)
Time Frame: Measured at week 1 and 26
Population: Participants in each group
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 19 | 19
Participants
  Week 1 | 10 | 7
  Week 26 | 7 | 6

10. Secondary Outcome: Proportion of Participants in Each Group Who Report One or More Safer Sex Acts in Last Week
Description: Proportion of participants in each group who report one or more safer sex acts in last week (description)
Time Frame: as for outcome 4
Population: as for outcome 8
Arm/Group | All Participants
Number analyzed (Participants) | 0

11. Secondary Outcome: Proportion of Participants in Each Group Who Report One or More Safer Sex Acts in Last Month
Description: Proportion of participants in each group who report one or more safer sex acts in last month (description)
Time Frame: Measured at week 1 and 26
Population: Participants in each group
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 19 | 19
Participants
  Week 1 | 16 | 15
  Week 26 | 10 | 13

12. Secondary Outcome: Proportion of Participants in Each Group Who Report One or More HIV Preventive Care-seeking or Information-seeking Acts in Last Week
Description: Proportion of participants in each group who report one or more HIV preventive care-seeking or information-seeking acts in last week (description)
Time Frame: as for outcome 4
Population: as for outcome 8
Arm/Group | All Participants
Number analyzed (Participants) | 0

13. Secondary Outcome: Proportion of Participants in Each Group Who Report One or More HIV Preventive Care-seeking or Information-seeking Acts in Last Month
Description: Proportion of participants in each group who report one or more HIV preventive care-seeking or information-seeking acts in last month (description)
Time Frame: Measured at week 1 and 26
Population: Participants in each group
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 19 | 19
Participants
  Week 1 | 18 | 18
  Week 26 | 19 | 14

14. Secondary Outcome: Proportion of Participants in Each Group Who Report One or More Paid Hours of Work in the Last Week
Description: Proportion of participants in each group who report one or more paid hours of work in the last week (description)
Time Frame: as for outcome 4
Population: as for outcome 8
Arm/Group | All Participants
Number analyzed (Participants) | 0

15. Secondary Outcome: Proportion of Participants in Each Group Who Report One or More Paid Hours of Work in the Last Month
Description: Proportion of participants in each group who report one or more paid hours of work in the last month (description)
Time Frame: Measured weekly at week 1 and 26
Population: Participants in each group
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 19 | 19
Participants
  Week 1 | 6 | 7
  Week 26: number analyzed (Participants) | 18 | 19
  Week 26 | 15 | 9

ADVERSE EVENTS:
Time Frame: 20 weeks
Description: The study used a structured weekly participant checklist to document whether each participant experienced an intervention-related adverse event.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19

LIMITATIONS AND CAVEATS:
All measures were self-reported and may be subject to reporting biases.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-23): https://cdn.clinicaltrials.gov/large-docs/65/NCT03766165/Prot_SAP_000.pdf